CLINICAL TRIAL: NCT00427817
Title: PRO-STATE: Prognostic Interest of Serum Protein Profiles of Patients Undergoing a Prostate Biopsy: Search for a Profile Corresponding to Fast-developing Lesions and Characterization of Implicated Proteins.
Brief Title: PRO-STATE:Search for a Protein Profile Corresponding to Fast-developing Lesions and Characterization of Implicated Proteins in Prostate Carcinoma
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: DCIC 06 11
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Adenoma, Prostatic
Keywords: Adenoma, Prostatic; Prostate; Proteomics; Urology
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The main objective of this study is to realise serum protein profiles for each patient undergoing a prostate biopsy and to identify relevant proteins.

DETAILED DESCRIPTION:
In men, prostate carcinoma is the first cancer and the second cause of death by cancer. It is a slowly evolving disease with no prognostic marker of poor outcome.

Currently, the Prostate Specific Antigen (PSA) is the only available biological marker. It is a tissue marker and not a tumoral pathology control.

This is why new tissue markers are urgently needed to select patients with unfavourable evolution, in order to treat them rapidly by more effective methods such as chemotherapy, hormonotherapy or radiotherapy. This could improve survival time and quality of life.

Proteomic and clinical data comparison could point to new relevant molecules and permit the development of new biological tests for routine use.

SELDI-TOF-MS (Surface Enhanced Laser Desorption/Ionisation Mass Spectrometry) permits an extremely sensitive analysis of proteins. This method has been substantially ratified by the literature and a number of markers have already been identified, particularly for several cancer pathologies.

As far as prostate carcinomas are concerned, previous proteomic researches on serum have led to diagnostic parameters, differentiating healthy patients, patients with benign lesion and patients having malignant lesions. However, at present, no relevant protein has been identified. Moreover, no study has been carried out to characterize fast-developing lesions, in order to anticipate response to treatments.

The main objective of this study is to realise serum protein profiles for each patient undergoing a prostate biopsy and to identify relevant proteins.

The main judgement criteria will be intensity peaks in the protein profile (area and height) with reference to combined criteria (PSA rate, clinical stage, Gleason score).

Two groups will be compared:

* Group 1: Control (negative biopsy).
* Group 2: Prostate carcinoma (positive biopsy).

This group will be subdivided:

* Group 2a : favourable prognostic according to AMICO classification
* Group 2b : intermediate or unfavourable prognostic according to AMICO classification

This will contribute to setting up an aftercare database combining clinical data with biological data and protein profile.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing a prostate biopsy or a prostatectomy(according to common criteria).

Exclusion criteria:

* Patient refusing to take part in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing a prostate biopsy or a prostatectomy(according to common criteria).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Luc DESCOTES, MD, Principal Investigator — 14th floor D, Urology Department
Locations (1):
- Urology Department - University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Stattin P, Hakama M. Correspondence re: B-L. Adam et al., Serum protein fingerprinting coupled with a pattern-matching algorithm distinguishes prostate cancer from benign prostate hyperplasia and healthy men. Cancer Res., 62: 3609-3614, 2002. Cancer Res. 2003 May 15;63(10):2701; author reply 2701-2. No abstract available. PMID 12750300
- [Background] Conrads TP, Fusaro VA, Ross S, Johann D, Rajapakse V, Hitt BA, Steinberg SM, Kohn EC, Fishman DA, Whitely G, Barrett JC, Liotta LA, Petricoin EF 3rd, Veenstra TD. High-resolution serum proteomic features for ovarian cancer detection. Endocr Relat Cancer. 2004 Jun;11(2):163-78. doi: 10.1677/erc.0.0110163. PMID 15163296
- [Background] Lehrer S, Roboz J, Ding H, Zhao S, Diamond EJ, Holland JF, Stone NN, Droller MJ, Stock RG. Putative protein markers in the sera of men with prostatic neoplasms. BJU Int. 2003 Aug;92(3):223-5. doi: 10.1046/j.1464-410x.2003.04341.x. PMID 12887471
- [Background] Ornstein DK, Rayford W, Fusaro VA, Conrads TP, Ross SJ, Hitt BA, Wiggins WW, Veenstra TD, Liotta LA, Petricoin EF 3rd. Serum proteomic profiling can discriminate prostate cancer from benign prostates in men with total prostate specific antigen levels between 2.5 and 15.0 ng/ml. J Urol. 2004 Oct;172(4 Pt 1):1302-5. doi: 10.1097/01.ju.0000139572.88463.39. PMID 15371828
- [Background] Petricoin EF, Ardekani AM, Hitt BA, Levine PJ, Fusaro VA, Steinberg SM, Mills GB, Simone C, Fishman DA, Kohn EC, Liotta LA. Use of proteomic patterns in serum to identify ovarian cancer. Lancet. 2002 Feb 16;359(9306):572-7. doi: 10.1016/S0140-6736(02)07746-2. PMID 11867112
- [Background] Petricoin EF 3rd, Ornstein DK, Paweletz CP, Ardekani A, Hackett PS, Hitt BA, Velassco A, Trucco C, Wiegand L, Wood K, Simone CB, Levine PJ, Linehan WM, Emmert-Buck MR, Steinberg SM, Kohn EC, Liotta LA. Serum proteomic patterns for detection of prostate cancer. J Natl Cancer Inst. 2002 Oct 16;94(20):1576-8. doi: 10.1093/jnci/94.20.1576. PMID 12381711
- [Background] Xiao Z, Prieto D, Conrads TP, Veenstra TD, Issaq HJ. Proteomic patterns: their potential for disease diagnosis. Mol Cell Endocrinol. 2005 Jan 31;230(1-2):95-106. doi: 10.1016/j.mce.2004.10.010. PMID 15664456
- [Background] Ye B, Cramer DW, Skates SJ, Gygi SP, Pratomo V, Fu L, Horick NK, Licklider LJ, Schorge JO, Berkowitz RS, Mok SC. Haptoglobin-alpha subunit as potential serum biomarker in ovarian cancer: identification and characterization using proteomic profiling and mass spectrometry. Clin Cancer Res. 2003 Aug 1;9(8):2904-11. PMID 12912935
- [Background] Zhang Z, Bast RC Jr, Yu Y, Li J, Sokoll LJ, Rai AJ, Rosenzweig JM, Cameron B, Wang YY, Meng XY, Berchuck A, Van Haaften-Day C, Hacker NF, de Bruijn HW, van der Zee AG, Jacobs IJ, Fung ET, Chan DW. Three biomarkers identified from serum proteomic analysis for the detection of early stage ovarian cancer. Cancer Res. 2004 Aug 15;64(16):5882-90. doi: 10.1158/0008-5472.CAN-04-0746. PMID 15313933